CLINICAL TRIAL: NCT03487406
Title: Anti-platelet Therapy in the Primary Prevention of Cardiovascular Disease in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Anti-platelet Therapy in the Prevention of Cardiovascular Disease in Patients With COPD (APPLE-COPD: ICON 2)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Newcastle-upon-Tyne Hospitals NHS Trust (Other)
Collaborators: AstraZeneca (Industry); Newcastle University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 2014-005475-86
Record Dates: First submitted 2015-10-06; First posted 2018-04-04 (Actual); Last update posted 2018-04-04 (Actual); Status verified 2018-03

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Ticagrelor; Aspirin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo Ticagrelor & placebo Aspirin (Placebo Comparator): Placebo Ticagrelor 90 mg- one tablet, twice daily. Placebo Aspirin 75 mg- one tablet, once a day.
  Interventions: Drug: Placebo Aspirin; Drug: Placebo Ticagrelor
- Aspirin & Placebo Ticagrelor (Active Comparator): Aspirin 75mg - one tablet, once a day. Placebo Ticagrelor 90 mg- one tablet, twice daily.
  Interventions: Drug: Aspirin; Drug: Placebo Ticagrelor
- Placebo Aspirin & Ticagrelor (Active Comparator): Placebo Aspirin 75 mg - one tablet, once a day. Ticagrelor 90 mg- one tablet, twice daily.
  Interventions: Drug: Ticagrelor; Drug: Placebo Aspirin
- Aspirin & Ticagrelor (Experimental): Aspirin 75 mg - one tablet, once a day. Ticagrelor 90 mg- one tablet, twice daily.
  Interventions: Drug: Ticagrelor; Drug: Aspirin

INTERVENTIONS:
Drug: Ticagrelor — One 90 mg tablet, oral, twice daily for 6 months.
  Other Names: Brilique
  Arms: Aspirin & Ticagrelor; Placebo Aspirin & Ticagrelor
Drug: Aspirin — One 75 mg tablet, oral, once a day, for 6 months.
  Arms: Aspirin & Placebo Ticagrelor; Aspirin & Ticagrelor
Drug: Placebo Aspirin — Sugar tablet to mimic Aspirin 75 mg tablet One 75 mg tablet, oral, once a day, for 6 months.
  Arms: Placebo Aspirin & Ticagrelor; Placebo Ticagrelor & placebo Aspirin
Drug: Placebo Ticagrelor — Sugar tablet to mimic Ticagrelor 90 mg tablet. Once 90 mg tablet, oral, twice daily for 6 months.
  Arms: Aspirin & Placebo Ticagrelor; Placebo Ticagrelor & placebo Aspirin

SUMMARY:
Patients with COPD (chronic bronchitis and/or emphysema) are known to be at an increased risk of heart disease and death due to heart attacks. There are several possible reasons for this, one of which is an increased tendency of the blood to clot, that can give rise to blood clot formation in the coronary arteries, and lead to heart attack. Medications such as Aspirin and another new blood thinning tablet called Ticagrelor are already used for patients with heart attacks. Given that patients with COPD are at higher risk of heart attack, the investigators wish to see if these tablets that can prevent blood clot formation in heart arteries might also prevent heart attacks happening in COPD patients. The investigators hope to understand the effects by measuring clotting and inflammation in the blood. All patients will be followed up for 6-months.

In addition the investigators wish to study COPD patients who do not have a high risk of developing future heart problems using the QRISK score to study their well being over a 1 year period to see if they might also benefit from blood thinning medications.

DETAILED DESCRIPTION:
The APPLE-COPD: ICON2 trial is a double blinded, proof-of-concept, randomised controlled trial that will include patients who have not been previously targeted in clinical cardiovascular research. The study will consist of patients with a lung condition called chronic obstructive pulmonary disease (COPD) who have not previously been diagnosed with coronary artery disease (CAD) and yet are at higher risk of CAD, myocardial infarction, and excess mortality (as determined by QRISK2 score). The QRISK2 is a simple questionnaire for heart disease that uses well known risk factors such as age, high blood pressure, smoking status and abnormal cholesterol levels. A QRISK score over 20 (20% risk of a cardiovascular event over the next ten years) is already used as a prompt to consider cholesterol lowering therapy (such as statins).

Patients with COPD (chronic bronchitis and/or emphysema) are known to be at an increased risk of heart disease and death due to heart attacks. There are several possible reasons for this, one of which is an increased tendency of the blood to clot which can give rise to blood clot formation in the coronary arteries, and lead to heart attack. Medications such as Aspirin and another new blood thinning tablet called Ticagrelor are already used for patients with heart attacks. Given that patients with COPD are at higher risk of heart attack, the investigators wish to see if these tablets that can prevent blood clot formation in heart arteries, might also prevent heart attacks happening in COPD patients. The investigators hope to understand the effects by measuring clotting and inflammation in the blood.

Aspirin and Ticagrelor are widely used in the UK for the management of coronary artery disease. For purposes of this study, Aspirin and Ticagrelor will be treated as an Investigational Medicinal Product (IMP). As a 2x2 factorial design, the primary analyses are based on a comparison of i) Aspirin vs no Aspirin and ii) Ticagrelor vs. no Ticagrelor (resulting in 4 treatment arms). Treatment allocation will be blinded to both the investigator and the participant.

Participants allocated to the treatment arms will be requested to take their trial medication for 6 months and will then be followed up clinically for a further 6 months by the research team to monitor any adverse events and the participant's well-being.

Participants allocated to the observational arm will be followed up for 1 year.

At 1 year all trial procedures will end and the patient will continue to receive routine care by the clinical care team.

ELIGIBILITY:
Inclusion Criteria:

* Abnormal spirometry with FEV1<80% and FEV1/FVC ratio <70% of predicted
* Smoking history that is 10-pack years or greater (current or ex smokers can be included)
* Have capacity to consent

Exclusion Criteria:

* Any condition that is being concurrently treated through anticoagulation or antiplatelet therapy including Aspirin (any form of Aspirin) or Ticagrelor (atrial fibrillation, deep vein thrombosis, valve prosthesis, recent myocardial infarction, use of drug eluting stents)
* Other specific contraindications to management with antiplatelet medication (bleeding risks, allergies)
* Any contraindication for Aspirin and Ticagrelor use
* Other concurrent terminal illnesses with life expectancy less than 1 year (congestive cardiac failure, carcinoma etc)
* Current involvement in another clinical trial or exposure to another IMP within the previous 30 days
* COPD with an atypical cause (e.g. A1- antitrypsin deficiency)
* Patients who are unable to provide informed consent
* Planned/ Expected major surgery where anti-platelet therapy would be ceased
* Pregnancy, planned pregnancy or current breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2015-09; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Change in baseline ASPI and ADP-induced platelet aggregation at 6 months | Baseline to 6 months
  The primary outcome measure is platelet reactivity measured at 6-months. Response is calculated according to high platelet reactivity (HPR).
  Rates of HPR will be determined according to recently published definitions of HPR for multiple electrode aggregometry in patients undergoing percutaneous coronary intervention, >46 AU for ADP test and >40 for ASPI test. Response rate will be calculated on an intention to treat basis as the total number of patients responding as a proportion of all patients randomised and reported descriptively with 95% confidence intervals. Any patients who are not assessable at 6-months will be classed as a non-responder.

SECONDARY OUTCOMES:
Change in inflammatory markers (myeloperoxidase (MPO) measured by routine blood test at baseline, 1 month and 6 months | Baseline to 6 months
  Measuring changes in inflammatory markers to investigate if treatment with APT is associated with reduced inflammatory marker levels (myeloperoxidase (MPO)).
Change in inflammatory markers (interleukin-6 (IL-6) measured by routine blood test at baseline, 1 month and 6 months | Baseline to 6 months
  Measuring changes in inflammatory markers to investigate if treatment with APT is associated with reduced inflammatory marker levels (interleukin-6 (IL-6)).
Change in inflammatory markers (fibrinogen) measured by routine blood test at baseline, 1 month and 6 months | Baseline to 6 months
  Measuring changes in inflammatory markers to investigate if treatment with APT is associated with reduced inflammatory marker levels (fibrinogen).
Change in inflammatory markers (high sensitive C reactive protein (hsCRP) measured by routine blood test at baseline, 1 month and 6 months | Baseline to 6 months
  Measuring changes in inflammatory markers to investigate if treatment with APT is associated with reduced inflammatory marker levels (high sensitive C reactive protein (hsCRP)).
Change in inflammatory markers (tumor necrosis factor alpha (TNF) measured by routine blood test at baseline, 1 month and 6 months | Baseline to 6 months
  Measuring changes in inflammatory markers to investigate if treatment with APT is associated with reduced inflammatory marker levels (tumor necrosis factor alpha (TNF)).
Changes in carotid intima media thickness | Baseline to 6 months
  Carotid intima media thickness measured by an ultrasound scan
Changes in vascular stiffness (m/s) | Baseline and 6-months
  Changes in vascular stiffness as measured by a cuff (Meter/Second)
Quality of life using EuroQoL-5D-5L health-related quality of life instrument | Baseline and 6-months
  The EQ-5D-5L consists of the EQ-5D-5L descriptive system and the EQ Visual Analogue scale (EQ VAS). The descriptive system has 5 dimensions (mobility, self care, usual activities, pain/discomfort, anxiety/depression), each with 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. The respondent indicates his/her health state in each of the 5 dimensions. This decision results in a 1-digit number expressing the level selected for that dimension. The digits for 5 dimensions can be combined in a 5-digit number describing the respondent's health state. The EQ Visual Analogue Scale records the respondent's self-rated health on a vertical, visual analogue scale (0-100) where the endpoints are labelled 'Best imaginable health state' (100) and 'Worst imaginable health state' (0). This information will be used as a quantitative measure of health outcome as judged by the individual respondents.
St George's Respiratory Questionnaire for Chronic Obstructive Pulmonary Disease Patients (SGRQ-C) | Baseline and 6-months
  The SGRQ measures health impairment in patients with asthma and COPD. Scored 0-100 (with 0 = best outcome and 100 worst outcome)

OTHER OUTCOMES:
Rates of major and minor bleeding as defined by the TIMI scale | Baseline to 6 months
  Rates of bleeding will be classified as per the TIMI Scale:
  Major - Intracranial haemorrhage or a ≥5 g/dl decrease in the haemoglobin concentration or a ≥15% absolute decrease in the haematocrit Minor- Observed blood loss: ≥3 g/dl decrease in the haemoglobin concentration or ≥10% decrease in the haematocrit Minor- No observed blood loss: ≥4 g/dl decrease in the haemoglobin concentration or ≥12% decrease in the haematocrit Minimal- Any clinically overt sign of haemorrhage (including imaging) that is associated with a <3 g/dl decrease in the haemoglobin concentration or <9% decrease in the haematocrit All Adverse Events (AE) will be reported descriptively as the number of patients experiencing an AE as a proportion of the total number of patients starting treatment.
Rates of major and minor bleeding as defined by the Bleeding Academic Research Consortium (BARC) definition. | Baseline to 6 months
  Rates of bleeding will be defined by bleeding type i.e. Type 0 -Type 5b
Response on spirometry using the MRC dyspnoea scale (Breathlessness) | Baseline to 6 months
  Spirometry will be measured using the MRC Breathlessness Scale-
  1. - Not troubled by breathlessness except on strenuous exercise
  2. - Short of breath when hurrying or walking up a slight hill
  3. - Walks slower than contemporaries on the level because of breathlessness, or has to stop for breath when walking at own pace
  4. - Stops for breath after about 100 m or after a few minutes on the level
  5. - Too breathless to leave the house, or breathless when dressing or undressing
Forced Expiratory Volume (FEV1) and Forced Vital Capacity (FVC) measured by spirometry | Baseline to 6 months
  A spirometer will be used to measure Forced Expiratory Volume (FEV1) and Forced Vital Capacity (FVC).

CONTACTS AND LOCATIONS:
Overall Officials: Vijay Kunadian, MBBS MD FRCP, Principal Investigator — Intitute of Cellular Medicine, Newcastle University
Locations (1):
- Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne, United Kingdom